CLINICAL TRIAL: NCT04396223
Title: TROPHAMET, a Phase I/II Trial of Avelumab and METhotrexate in Low-risk Gestational TROPHoblastic Neoplasias as First Line Treatment
Brief Title: Avelumab and Methotrexate in in Low-risk Gestational Trophoblastic Neoplasias as First Line Treatment
Acronym: TROPHAMET
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18 0857
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Gestational Trophoblastic Neoplasias (GTN)
Keywords: avelumab; methotrexate; PDL1; gestational trophoblastic neoplasias, GTN; hydatiform mole; hCG,
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab combined with methotrexate and folinic acid (Experimental): Avelumab administration at 800 mg every 2 weeks and methotrexate administration at 1mg/kg/day during 4 months ½ (median)
  Interventions: Drug: Avelumab Injection; Drug: Methotrexate 1 GM Injection

INTERVENTIONS:
Drug: Avelumab Injection — Avelumab administration at 800mg a 1 hour IV infusion once every 14 days during 4 months ½ (median)
Drug: Methotrexate 1 GM Injection — methotrexate administration at 1mg/kg/day during 4 months ½ (median)

SUMMARY:
Gestational trophoblastic neoplasias (GTN) are characterized by the persistence of elevated hCG titers after complete uterine evacuation of a partial hydatidiform mole (PHM) or a complete hydatidiform mole.

Low-risk GTN patients (FIGO score ≤ 6) are commonly treated with single agent treatment (methotrexate or actinomycin-D) The cure rate, assessed by hCG normalization, is obtained in 65 to 75% of patients with these agents GTN patients with resistance to these treatments are treated with another single agent drug or polychemotherapy regimens, such as EMA-CO or BEP regimen.

Chemotherapy standard regimens are old and toxic for these young lady patients, with potential long term effects detrimental for further maternity and quality of life

There is a strong rational for investigating the anti-PDL1 monoclonal antibody avelumab in chemoresistant GTN patients. Several elements suggest that the normal pregnancy immune tolerance is "hijacked" by GTN cell for proliferating :

* Spontaneous regressions of metastastic GTN are regularly observed, thereby the role of immune system for rejecting GTN cells.
* Strong and constant overexpression of PDL1 and NK cells has been found in all subtypes and settings of GTN tumors from French reference gestational trophoblastic center.
* Complete and durable responses to pembrolizumab were reported in 3 patients with multi-chemoresistant GTN in United Kingdom.
* Three cases of hCG normalization with avelumab in 6 patients with chemo-resistant GTN enrolled in TROPHIMMUN cohort A (resistant to a mono-chemotherapy).
* Cytotoxicity of avelumab is mediated through antibody dependent cell cytotoxicity (ADCC) by NK cells.

ELIGIBILITY:
Inclusion Criteria:

* - Woman older than 18 years
* Low-risk gestational trophoblastic neoplasia according to FIGO score (FIGO score ≤ 6) with indication of methotrexate as first line treatment
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients with adequate bone marrow function measured within 28 days prior to administration of study treatment as defined below

  * Absolute granulocyte count ≥ 1.5 x 10 9 /L
  * Platelet count ≥ 100 x 10 9 /L
  * Haemoglobin ≥ 9.0 g/dL (may have been blood transfused)
* Patients with adequate renal function:

  * Calculated creatinine clearance ≥ 30 ml/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Patients with adequate hepatic function

  *Serum bilirubin ≤ 1.5 x UNL and AST/ALT ≤ 2.5 X UNL (≤ 5 X UNL for patients with liver metastases)
* Patients must have a life expectancy ≥ 16 weeks
* Confirmation of non-childbearing status for women of childbearing potential.

An evolutive pregnancy can be ruled out in the following cases:

* in case of a previous hysterectomy
* if serum hCG level ≥ 2 000 IU/L and no intra or extra-uterine gestational sac is detected on pelvic ultrasound
* if serum hCG level < 2 000 IU/L on a first measurement and serum hCG increases <100% on a second measurement performed 3 days later.

  * Highly effective contraception if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential must agree to use 2 highly effective contraceptions, defined as methods with a failure rate of less than 1 % per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 12 months after avelumab treatment.
  * Patients who gave its written informed consent to participate to the study
  * Patients affiliated to a social insurance regime
  * Patient is willing and able to comply with the protocol for the duration of the treatment

Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- CTLA 4 antibody (including ipilimumab, tremelimumab or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways).
* Illness, incompatible with avelumab, such as congestive heart failure; respiratory distress; liver failure; uncontrolled epilepsy; allergy.
* Patients with a known allergic hypersensitivity to methotrexate or any of the other ingredients (sodium chloride, sodium hydroxide, and hydrochloric acid if excipient)
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* All subjects with brain metastases, except those meeting the following criteria:

  * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrolment, No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable).
  * Subjects with brain metastases must be either off steroids except a stable or decreasing dose of <10mg daily prednisone (or equivalent).
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
* Persistent toxicities (>=CTCAE grade 2) with the exception of alopecia and sensory neuropathy, caused by previous cancer therapy.
* Treatment with other investigational agents.
* Bowel occlusive syndrome, inflammatory bowel disease, immune colitis, or other gastro-intestinal disorder that does not allow oral medication such as malabsorption.
* Stomatitis, ulcers of the oral cavity and known active gastrointestinal ulcer disease
* Clinically significant (i.e., active) and severe cardiovascular disease according to investigator opinion such as myocardial infarction (< 6 months prior to enrollment)
* Patients with immune pneumonitis, pulmonary fibrosis
* Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of partially controlled asthma Global Initiative for Asthma 2011).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
* Active infection requiring systemic therapy.
* Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
* Administration of a live vaccine within 30 days prior to study entry.
* Current or prior use of immunosuppressive medication within 7 days prior to start of study treatment.

The following are exceptions to this exclusion criterion:

* Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection);
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent;
* Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).

  * Active autoimmune disease that might deteriorate when receiving an immunostimulatory agents.

Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.

* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control.
* Treatment with oral anticoagulant such Coumadin.
* Alcoholism (patient interview, investigator judgment)
* Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome. Torsades de Pointes, arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation, bradycardia defined as <50 bpm), right bundle branch block and left anterior hemiblock (bifascicular block), unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF New York Heart Association Class III or IV), cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
* Prior organ transplantation, including allogeneic stem cell transplantation (excluding autologous bone marrow transplant)
* Patients under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2025-04-12 (Estimated); Study Completion 2028-10-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities of methotrexate and avelumab combination in low-risk GTN patients as first line. | treatment duration 3 months (median estimation)
  Safety run-in: dose-limiting toxicities (DLT) will be determined during the first 3 months after the start of treatment
Rate of patients with successful normalization of hCG | treatment duration 3 months (median estimation)
  The main endpoint of this study is the rate of patients with successful normalization of hCG allowing for treatment discontinuation (hCG normalization). Patients will continue on treatment until the weekly hCG assays reach the institutional normal threshold, and then for 3 additional cycles, or otherwise will be stopped in the case of resistance, defined as a rise (a > 20% rise between two assays, observed twice on three consecutive weekly assays) or a plateau (a < 10% decrease between two assays observed three times on four consecutive weekly assays) in the hCG level, or unacceptable toxicity and/or death.

SECONDARY OUTCOMES:
Evaluate the safety of methotrexate and avelumab combination administration | during treatment duration (3 months), 1 month after end of treatment and 36 months after end of treatment (median : 8 months 1/2).
  To assess the rate of treatment-emergent adverse events (TEAEs) and treatment-related adverse events (AEs), treatment-related Grade ≥ 3 AEs, and immune-related AEs, according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)
To assess the efficacy of avelumab and methotrexate in terms of resistance-free survival in low-risk GTN patients as first line setting | during treatment (3 months median), 1 month after the end of treatment and 36 months after the end of treatment
  Resistance rate will be evaluated according to hCG level.
To assess the efficacy of avelumab and methotrexate in terms of resistance-free survival in low-risk GTN patients as first line setting | during treatment (3 months median), 1 month after the end of treatment and 36 months after the end of treatment
  Resistance-free survival will be evaluated according to hCG level.
To assess the efficacy of avelumab and methotrexate in terms of relapse free survival in low-risk GTN patients as first line setting after an initial hCG normalization that enabled study treatment discontinuation | during treatment (3 months median), 1 month after the end of treatment and 36 months after the end of treatment
  Relapse-free survival will be evaluated in the case of relapse requiring treatment resumption after a hCG normalization that enabled study treatment discontinuation
To assess the efficacy of avelumab and methotrexate in terms of overall survival in low-risk GTN patients as first line setting | during treatment (3 months median), 1 month after end of treatment and 36 months after end of treatment
  Overall survival

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Pierre Bénite
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Assistance Publique Hôpitaux de Paris, Paris
  - Centre Eugène Marquis, Rennes
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse